CLINICAL TRIAL: NCT05453097
Title: Prognostic Value of the Selvester QRS Score for Perioperative Myocardial Injury Following Non-cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Deniz Mutlu, Fellow, Istanbul University - Cerrahpasa
Other Study IDs: 2022/172
Record Dates: First submitted 2022-06-26; First posted 2022-07-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Ischemia; Cardiac Arrhythmia; Perioperative Injury; Perioperative Complication
Keywords: myocardial injury; Perioperative injury
MeSH Terms: conditions — Coronary Artery Disease; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cardiac Troponin and routine biochemical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perioperative Myocardial Injury Occured: Patients with troponin elevation from the preoperative basal level do not meet the criteria for myocardial infarction according to the fourth universal myocardial infarction guideline, do not describe active anginal complaints, and underwent surgery in the operating room.
  Interventions: Diagnostic Test: Selvester QRS Score with Preoperative ECG
- Perioperative Myocardial Injury Not Occured: Patients without troponin elevation from the preoperative basal level, do not describe active anginal complaints, and underwent surgery in the operating room.
  Interventions: Diagnostic Test: Selvester QRS Score with Preoperative ECG

INTERVENTIONS:
Diagnostic Test: Selvester QRS Score with Preoperative ECG — Selvester QRS score will be calculated with the preoperative ECG of the patients.

SUMMARY:
The purpose of this study to determine the prognostic value of the Selvester QRS score for perioperative myocardial injury following elective non-cardiac surgery.

DETAILED DESCRIPTION:
This study was designed as an investigator-directed, non-commercial, observational, prospective, national, single-center study. The effect of preoperative complex ECG changes on the formation of cardiac damage will be studied. The data of the people participating in the study will be kept entirely confidential. After being informed about the study, all patients giving written informed consent will undergo preoperative evaluation. An ECG and cardiac troponin analysis will be performed to the patients who meet the eligibility. After the surgery will be completed control cardiac troponin and extensive physical examination will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergoing elective non-cardiac surgery in the operating room
* ≥18 years old
* Interpretable preoperative ECG of the patient
* Preoperative negative high sensitive Cardiac Troponin T
* ASA I-III class
* Patients who give the informed consent

Exclusion Criteria:

* A history of myocardial infarction, coronary artery disease, PCI and revascularization
* A history of chronic renal disease, cerebrovascular incident, stroke
* ASA class IV
* Patients who do not give the informed consent
* Patients who undergoing emergency surgery
* Patients whose preoperative ECG is not interpretable
* Minor procedures to be performed outside or inside the operating room

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on patients aged 18-90 years who have had elective surgery (besides cardiac operations) performed by a surgeon in the operating rooms of a tertiary university hospital, whose ECG before the operation is interpretable, and whose troponin value is measured before and after the operation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The prediction of perioperative cardiac injury with preoperative Selvester ECG Score | Change from Baseline cardiac troponin levels at postoperative 1st hour in PACU
  Selvester ECG score is a validated technique for predicting myocardial scar and injury level in patients who undergone PCI. It is aimed to predict and demonstrate perioperative myocardial damage using this algorithm.

SECONDARY OUTCOMES:
The prediction of preoperative high-sensitivity troponin and ECG abnormalities on arrhythmia susceptibility. | Arrhythmia surveillance during peroperative and postoperative 1st hour in PACU
  The prediction of preoperative high-sensitivity troponin and ECG abnormalities on arrhythmia susceptibility by monitoring the cardiac rhythm
Effect of preoperative cardiac assessment on postoperative cardiac adverse event | Cardiac adverse event surveillance during peroperative and postoperative 24 hours
  Effect of preoperative cardiac assessment on postoperative cardiac adverse event
Determination of postoperative intensive care hospitalizations for cardiac reasons | postoperative intensive care hospitalizations for cardiac reasons until postoperative 24 hours
  Determination of the reasons of the postoperative intensive care unit hospitalizations for cardiac reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Kivanc Yalin, MD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Loring Z, Chelliah S, Selvester RH, Wagner G, Strauss DG. A detailed guide for quantification of myocardial scar with the Selvester QRS score in the presence of electrocardiogram confounders. J Electrocardiol. 2011 Sep-Oct;44(5):544-54. doi: 10.1016/j.jelectrocard.2011.06.008. PMID 21872001
- [Result] Sapra R, Hallqvist L, Schlegel TT, Ugander M, Bell M, Maanja M. Predicting peri-operative troponin elevation by advanced electrocardiography. J Electrocardiol. 2021 Sep-Oct;68:1-5. doi: 10.1016/j.jelectrocard.2021.06.008. Epub 2021 Jul 2. PMID 34246860